CLINICAL TRIAL: NCT05575323
Title: Stereotactic Body Radiotherapy and pedicLE Screw fixatioN During One Hospital Visit for Patients With Painful Unstable Spinal Metastases: A Randomized Trial (BLEND)
Brief Title: Randomized Trial on Same-day SBRT and Surgical Stabilization for Symptomatic Spinal Metastases
Acronym: BLEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Prof. H.M. Verkooijen, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80847.041.22
Record Dates: First submitted 2022-09-29; First posted 2022-10-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Spinal Metastases
Keywords: Spinal metastases; SBRT; Surgery; Same-day treatment; RCT
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Masking Description: According to the TwiCs design, patients allocated to the control group are not informed about their role as a control in the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients will receive high dose, single fraction stereotactic body radiotherapy (SBRT) using differential dosing: 18 or 21 Gy on the metastasis. Within 24 hours after SBRT, patients will have surgical stabilization with or without decompression.
  Interventions: Other: Same-day SBRT and spinal surgery
- Control (Active Comparator): Patients will undergo the standard of care, which is surgical stabilization with or without decompression, followed by conventional radiotherapy (cRT) or SBRT as soon as the wound is healed sufficiently.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Same-day SBRT and spinal surgery — SBRT and surgical stabilization with or without decompression within 24 hours
  Arms: Intervention
Other: Standard of care — Surgical stabilization with or without decompression followed by cRT or SBRT as soon as the wound is healed sufficiently
  Arms: Control

SUMMARY:
The BLEND RCT aims to evaluate the (cost-)effectiveness of same-day SBRT and surgical stabilization with or without decompression for the treatment of symptomatic, unstable spinal metastases on physical functioning four weeks after the start of treatment, compared with the standard of care (surgery followed by radiotherapy as soon as the wound healed sufficiently).

DETAILED DESCRIPTION:
Rationale: Currently, patients with unstable spinal metastases receive surgical stabilization with/without decompression followed by conventional radiotherapy (cRT) or stereotactic body radiotherapy (SBRT) as soon as wound healing allows (at least 1 week). Advancements in radiotherapy techniques makes preoperative radiotherapy possible with sparing of the soft tissues overlying the surgical field. This makes it possible to shorten or even eliminate the time interval between surgery and radiotherapy. This will result in shorter and less hospital visits, earlier pain relief from irradiation, and faster return to systemic therapy without an increase in wound complications due to the short interval between surgery and radiotherapy.

Objective: The BLEND RCT aims to evaluate the (cost-)effectiveness of same-day SBRT and surgery for the treatment of symptomatic, unstable spinal metastases on physical functioning four weeks after the start of the treatment, compared with the standard of care (surgery followed by radiotherapy, i.e., CRT or SBRT).

Study design: A phase II randomized controlled trial within the PRospective Evaluation of interventional StudiEs on boNe metastases (PRESENT) cohort including patients with bone metastases, according to the Trials within Cohorts (TwiCs) design.

Study population: Patients with symptomatic (cervical, thoracic and/or lumbar) spinal metastases and impending spinal instability requiring radiotherapy and surgical stabilization with or without decompression.

Intervention: SBRT (with active dose-sparing of the surgical site) and surgical stabilization with or without decompression within 24 hours. The control group will receive the standard of care, which is surgical stabilization with or without decompression followed by cRT or SBRT as soon as the wound is healed sufficiently.

Main study endpoints: The primary endpoint is physical functioning at four weeks after the start of the treatment. Secondary endpoints are pain response, duration of pain relief, length of hospital stay, time to return to systemic therapy, neurological deterioration, adverse events (e.g. wound complications), quality of life and survival. In addition, we will study the cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic (cervical, thoracic and/or lumbar) spinal metastases from solid tumors and (impending) spinal instability requiring radiotherapy and surgical decompression and/or stabilization
* Histologic proof of malignancy or radiographic/clinical characteristics indicating malignancy beyond reasonable doubt
* Radiographic evidence of spinal metastases
* Participation in PRESENT cohort, including consent for randomization into future trials
* Fit for (radio)surgery
* Age >18 years
* Written informed consent

Exclusion Criteria:

* SBRT cannot be delivered, e.g. in patients who cannot lie on the treatment table because of pain
* Routine surgical decompression and/or stabilization and radiotherapy cannot be performed, e.g., multiple spinal metastases requiring surgical bridging of more than five vertebral levels and/or requiring radiotherapy on more than one location
* Prior surgery or radiotherapy to the index level(s)
* Multiple myeloma
* Neurological deficits (ASIA C, B or A), or partial neurological deficits (ASIA D) with rapid progression (hours to days)
* Treated with Bevacizumab and other medication with long half-life that interferes with radiotherapy
* Life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical functioning | at 4 weeks after the start of treatment
  Physical functioning is a functional scale from the EORTC QLQ-C15-PAL questionnaire. Patients rate each item on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much), and scale scores were linearly transformed to a 0-100 scale. A higher score on the functional scale indicates better functioning.

SECONDARY OUTCOMES:
Pain response | at 2, 4, 6 and 8 weeks, and 3 months after the start of treatment
  Pain response is defined as 1) a decline in worst pain score of at least two points on an NRS of ten at the treated site without increase in analgesic use, or 2) an analgesic decrease of at least 25% without an increase in pain score. Worst pain score will be measured with the Brief Pain Inventory.
Duration of pain relief | up to 3 months
  Duration of pain relief as measured by the Brief Pain Inventory (BPI).
Duration of hospital stay | up to 3 months
  Duration of hospital stay in days
Days until return to systemic treatment | up to 12 months
  Days until return to systemic treatment
Neurological deterioration | up to 12 months
  Occurrence of neurological deterioration is defined as deterioration of more than one grade on the American Spinal Cord Injury Association (ASIA) scale as measured by physical examination by a neurologists or trained ASIA physician.
Change in health-related quality of life | at 4 and 8 weeks, and 3 and 6 months after the start of treatment
  Change in patient-reported health-related quality of life is measured by the EORTC QLQ-C15-PAL at predefined time intervals.
Change in health-related quality of life | at 4 and 8 weeks, and 3 and 6 months after the start of treatment
  Change in patient-reported health-related quality of life is measured by the EORTC QLQ-BM22 at predefined time intervals.
Local control | up to 12 months
  Local control according to routine imaging and electronic patient chart
Adverse events | up to 3 months
  Adverse events are defined as any undesirable experience occurring to a patient during the study, (likely) related to the experimental treatment procedure. All adverse events during hospital stay will be evaluated using the most recent version of the National Cancer Institute Common Toxicity Criteria of Adverse Events (CTCAE; version 5.0, version 6.0 when available at the start of the study) for acute and late toxicity. All adverse events after hospital discharge reported spontaneously by the patient or observed by the investigator or research team will be recorded up to three months after the treatments.
Progression free survival | up to 12 months
  Progression free survival is defined as time between treatment and first sign of progression of disease.
Overall survival | up to 12 months
  Overall survival is defined as time between treatment and death from any cause.

OTHER OUTCOMES:
Cost-effectiveness | up to 12 months
  If same-day SBRT and surgery is more costly and more effective than the standard of care, an incremental cost-effectiveness ratio (ICER) will be calculated by dividing the extra QALYs by the extra effects. This will give an estimation of the extra costs that are needed to gain one QALY. If this is below the cost-effectiveness threshold, same-day SBRT and surgery is deemed cost-effective. If either same-day SBRT and surgery or the standard of care is less costly and more effective than its alternative, it dominates this alternative and no ICER is necessary to determine cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Helena M. Verkooijen, Prof, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huele EH, van der Velden JM, Kasperts N, Eppinga WSC, Grutters JPC, Suelmann BBM, Weening AA, Delawi D, Teunissen SCCM, Verkooijen HM, Verlaan JJ, Gal R. Stereotactic Body radiotherapy and pedicLE screw fixatioN During one hospital visit for patients with symptomatic unstable spinal metastases: a randomized trial (BLEND RCT) using the Trials within Cohorts (TwiCs) design. Trials. 2023 May 4;24(1):307. doi: 10.1186/s13063-023-07315-y. PMID 37143158